CLINICAL TRIAL: NCT06611631
Title: Clinical and Radiographic Evaluation of Hyaluronic Acid (Gengigel Teething) Versus Mineral Trioxide Aggregate( Angelus) as Pulpotomy Agent in Vital Primary Molars: A Randomized Clinical Trial
Brief Title: Clinical and Radiographic Evaluation of Hyaluronic Acid (Gengigel Teething) Versus Mineral Trioxide Aggregate( Angelus) as Pulpotomy Agent in Vital Primary Molars
Acronym: HA - MTA
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hadeer Nasser Hammad Aboeldahb, Pediatric Resident, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HA Pulpotomy
Record Dates: First submitted 2024-09-22; First posted 2024-09-25 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-11

CONDITIONS: Pulpotomies Primary Teeth; Pulp Disease, Dental
Keywords: hyaluronic acid; HA; MTA; Mineral Trioxide Aggregate
MeSH Terms: conditions — Dental Pulp Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hyaluronic Acid Pulpotmoy (Experimental): 1. After complete hemostasis, pulp stumps will be covered with a mixture of Hyaluronic acid gel and zinc oxide powder to reach suitable consistency (1:1 ratio by volume) then gentle condensation in the pulp chamber will be done by a moistened cotton pellet and then the rest of the pulp chamber will be filled by glass ionomer restoration .
  2. Tooth will be restored with stainless steel crown.
  Interventions: Procedure: Hyaluronic acid pulpotomy
- Mineral Trioxide Aggregate (Active Comparator): 1. After complete hemostasis, MTA+ saline will be manipulated in the ratio of 3:1 (powder: liquid) to obtain a putty mix. This mix will be placed over the radicular pulp with the help of a suitable sterile amalgam carrier. Gentle condensation of the mix will be done in the pulp chamber with a moistened cotton pellet, followed by the application of glass ionomer restoration.
  2. Tooth will then be restored with stainless steel crown.
  Interventions: Procedure: mineral trioxide aggregate pulpotomy

INTERVENTIONS:
Procedure: Hyaluronic acid pulpotomy — 1. After complete hemostasis, pulp stumps will be covered with a mixture of Hyaluronic acid gel and zinc oxide powder to reach suitable consistency (1:1 ratio by volume) then gentle condensation in the pulp chamber will be done by a moistened cotton pellet and then the rest of the pulp chamber will be filled by glass ionomer restoration .
  2. Tooth will be restored with stainless steel crown.
  Other Names: HA pulpotomy
  Arms: Hyaluronic Acid Pulpotmoy
Procedure: mineral trioxide aggregate pulpotomy — 1. After complete hemostasis, MTA+ saline will be manipulated in the ratio of 3:1 (powder: liquid) to obtain a putty mix. This mix will be placed over the radicular pulp with the help of a suitable sterile amalgam carrier. Gentle condensation of the mix will be done in the pulp chamber with a moistened cotton pellet, followed by the application of glass ionomer restoration.
  2. Tooth will then be restored with stainless steel crown.
  Other Names: MTA pulpotomy
  Arms: Mineral Trioxide Aggregate

SUMMARY:
The goal of this clinical trial is to Clinical and Radiographic Evaluation of Hyaluronic Acid (Gengigel Teething) Versus Mineral Trioxide Aggregate( Angelus) as Pulpotomy Agent in Vital Primary Molars.

The main question it aims to answer is:

Is there a difference in the clinical or radiographic success when using Hyaluronic acid (Gengigel Teething, Ricerfarma , Italy) versus mineral trioxide aggregate (Angelus, Londrina ,Brazil) in pulpotomy of carious primary molars in children?

DETAILED DESCRIPTION:
Preservation of primary dentition decreases the risk of developing any occlusal abnormalities caused by premature loss of primary teeth, which are considered natural space maintainers for the successor permanent teeth, therefore vital pulp therapy is of a big concern in the research field in pediatric dentistry.

One of the most commonly used regenerative materials in pulpotomies is Mineral Trioxide Aggregate (MTA) which showed a high success rate clinically and radiographically when compared to other materials due to its biocompatibility, antibacterial properties and excellent sealing ability . However it has some drawbacks such as difficult manipulation and handling because it is supplied in powder and liquid form which need mixing. Mixing is operator dependent and may be not uniform if handled wrongly, technique sensitive, potential discoloration, and long setting time.

Hyaluronic acid have been introduced as a new biologically based therapeutics directed at preserving pulp vitality. Owing to good handling characteristics, biocompatibility, odontogenic property. non-toxic, biodegradable ,non-immunogenic , anti-inflammatory and antibacterial action, hyaluronic acid is a promising pulpotomy agent Furthermore, the use of a gel containing HA facilitated faster healing in laser-induced wounds by secondary intention. HA tends to be helpful in the treatment of swelling and trismus as well as the inflammatory reaction after third molar extraction.

The benefits of this study to the participants:

A cheaper , faster and easier clinical procedure leads to a more efficient dental treatment, which could develop positive attitude of children towards dentistry.

The benefits of this study to the population:

1. Providing better quality of dental treatment.
2. Enhance the overall oral health of children.

The benefits of this study to the clinicians:

1. Providing a new biological and alternative treatment option.
2. Decreased chairside time owing to its better manipulation and less technique sensitive .
3. cheaper and accessible alternative .

ELIGIBILITY:
Inclusion Criteria:

* Patients:

Aged 4-8 years, in good general health and medically within normal.

Teeth:

* Restorable mandibular primary molars.
* History of reversible pulpitis.

Pre-operative Radiographic criteria:

* Absence of periapical or inter-radicular radiolucencies.
* Absence of widening of periodontal ligaments (PDL) space.
* Absence of internal or external root resorption.

Exclusion Criteria:

Patients:

* With systemic disorders.
* Physical or mental disabilities.
* Unable to attend follow- up visits.
* Refusal of Participation.
* Refusal to sign the informed consent.

Teeth:

* Previously accessed teeth.
* Mobile mandibular primary molars.
* Swelling in the vestibule or on palpation.
* Pain on percussion

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Absence of post- operative pain. | 1 week changes from baseline pulp condition
  Asking the patient and/or guardian. Outcome measuring unit :Binary (present/absent)
Absence of pain on percussion. | at 3 month, change from the baseline pulp condition at 6 month, change from baseline pulp condition at 9 month, change from base line pulp condition at 12 month.
  Percussion test using the back of a dental mirror. Outcome measuring unit :Binary (present/absent)
Absence of Swelling. | at 3 month, change from the baseline pulp condition at 6 month, change from baseline pulp condition at 9 month, change from base line pulp condition at 12 month.
  Visual examination. Outcome measuring unit :Binary (present/absent)
Absence of Sinus or fistula. | at 3 month, change from the baseline pulp condition at 6 month, change from baseline pulp condition at 9 month, change from base line pulp condition at 12 month.
  Visual examination. Outcome measuring unit :Binary (present/absent)
Pathologic mobility | at 3 month, change from the baseline pulp condition at 6 month, change from baseline pulp condition at 9 month, change from base line pulp condition at 12 month.
  Mobility test (pressure using the end of two dental mirrors). Outcome measuring unit :Binary (present/absent)

SECONDARY OUTCOMES:
Absence of external or internal root resorption. | at 3 month, change from the baseline pulp condition at 6 month, change from base line pulp condition at 12 month.
  Intraoral digital periapical X-ray. Outcome measuring unit :Binary (present/absent)
Absence of furcation or periapical radiolucency. | at 3 month, change from the baseline pulp condition at 6 month, change from base line pulp condition at 12 month.
  Intraoral digital periapical X-ray. Outcome measuring unit :Binary (present/absent)
Absence of any adverse radiographic finding. | at 3 month, change from the baseline pulp condition at 6 month, change from base line pulp condition at 12 month.
  Intraoral digital periapical X-ray. Outcome measuring unit :Binary (present/absent)

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smail-Faugeron V, Fron Chabouis H, Durieux P, Attal JP, Muller-Bolla M, Courson F. Development of a core set of outcomes for randomized controlled trials with multiple outcomes--example of pulp treatments of primary teeth for extensive decay in children. PLoS One. 2013;8(1):e51908. doi: 10.1371/journal.pone.0051908. Epub 2013 Jan 3. PMID 23300955
- [Background] Chan AW, Pello A, Kitchen J, Axentiev A, Virtanen JI, Liu A, Hemminki E. Association of Trial Registration With Reporting of Primary Outcomes in Protocols and Publications. JAMA. 2017 Nov 7;318(17):1709-1711. doi: 10.1001/jama.2017.13001. PMID 28892118
- [Background] Higgins JPT, Thomas J, Chandler J, Cumpston M, Li T, Page MJ, Welch VA (editors). Cochrane Handbook for Systematic Reviews of Interventions version 6.3 (updated February 2022). Cochrane, 2022.
- [Background] Camilleri J. Hydration characteristics of Biodentine and Theracal used as pulp capping materials. Dent Mater. 2014 Jul;30(7):709-15. doi: 10.1016/j.dental.2014.03.012. Epub 2014 Apr 29. PMID 24793199
- [Background] Al-Johany SS, Al Amri MD, Alsaeed S, Alalola B. Dental Implant Length and Diameter: A Proposed Classification Scheme. J Prosthodont. 2017 Apr;26(3):252-260. doi: 10.1111/jopr.12517. Epub 2016 Jul 5. PMID 27379723
- [Background] Xu X, Jha AK, Duncan RL, Jia X. Heparin-decorated, hyaluronic acid-based hydrogel particles for the controlled release of bone morphogenetic protein 2. Acta Biomater. 2011 Aug;7(8):3050-9. doi: 10.1016/j.actbio.2011.04.018. Epub 2011 Apr 24. PMID 21550426
- [Background] Cowman MK, Lee HG, Schwertfeger KL, McCarthy JB, Turley EA. The Content and Size of Hyaluronan in Biological Fluids and Tissues. Front Immunol. 2015 Jun 2;6:261. doi: 10.3389/fimmu.2015.00261. eCollection 2015. PMID 26082778
- [Background] Koray M, Ofluoglu D, Onal EA, Ozgul M, Ersev H, Yaltirik M, Tanyeri H. Efficacy of hyaluronic acid spray on swelling, pain, and trismus after surgical extraction of impacted mandibular third molars. Int J Oral Maxillofac Surg. 2014 Nov;43(11):1399-403. doi: 10.1016/j.ijom.2014.05.003. Epub 2014 Jun 10. PMID 24924267
- [Background] Romeo U, Libotte F, Palaia G, Galanakis A, Gaimari G, Tenore G, Del Vecchio A, Polimeni A. Oral soft tissue wound healing after laser surgery with or without a pool of amino acids and sodium hyaluronate: a randomized clinical study. Photomed Laser Surg. 2014 Jan;32(1):10-6. doi: 10.1089/pho.2013.3509. Epub 2013 Dec 14. PMID 24328847
- [Background] Bagio DA, Lestari NA, Putra WA, Alinda SD, Ricardo S, Julianto I. The effect of hyaluronic acid conditioned media on hDPSCs differentiation through CD44 and transforming growth factor-beta1 expressions. J Adv Pharm Technol Res. 2023 Apr-Jun;14(2):89-93. doi: 10.4103/japtr.japtr_649_22. Epub 2023 Apr 13. PMID 37255878
- [Background] Motwani N, Ikhar A, Nikhade P, Chandak M, Rathi S, Dugar M, Rajnekar R. Premixed bioceramics: A novel pulp capping agent. J Conserv Dent. 2021 Mar-Apr;24(2):124-129. doi: 10.4103/JCD.JCD_202_20. Epub 2021 Oct 9. PMID 34759576
- [Background] Cordell S, Kratunova E, Marion I, Alrayyes S, Alapati SB. A Randomized Controlled Trial Comparing the Success of Mineral Trioxide Aggregate and Ferric Sulfate as Pulpotomy Medicaments for Primary Molars. J Dent Child (Chic). 2021 May 15;88(2):120-128. PMID 34321144
- [Background] Igna A. Vital Pulp Therapy in Primary Dentition: Pulpotomy-A 100-Year Challenge. Children (Basel). 2021 Sep 24;8(10):841. doi: 10.3390/children8100841. PMID 34682106
- [Background] Guagnano R, Romano F, Defabianis P. Evaluation of Biodentine in Pulpotomies of Primary Teeth with Different Stages of Root Resorption Using a Novel Composite Outcome Score. Materials (Basel). 2021 Apr 24;14(9):2179. doi: 10.3390/ma14092179. PMID 33923152